CLINICAL TRIAL: NCT00682955
Title: Comparing the Efficacy of Different Zinc Formulations in the Treatment of Acute Diarrhea Among Young Children at Hospital Based Setting in Pakistan
Brief Title: Comparing the Efficacy of Different Zinc Formulations in the Treatment of Diarrhea
Acronym: Zinc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Civil Hospital, Hyderabad, Pakistan (Unknown); National Institute of Child Health, Karachi, Pakistan (Other Government)
Responsible Party: Dr Zulfiqar A Bhutta, The Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 857-PED/ERC-07
Record Dates: First submitted 2008-05-20; First posted 2008-05-23 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Incidence of Acute Diarrhea; Incidence of Abdominal Pain
Keywords: Diarrhea; Zinc Sulphate; Efficacy
MeSH Terms: conditions — Diarrhea | interventions — Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Active Comparator): This group has been given Zinc Sulphate in Suspension Form.
  Interventions: Drug: Zinc Sulphate
- A (Active Comparator): This group has been given Tablets of Zinc Sulphate.
  Interventions: Drug: Zinc Sulphate

INTERVENTIONS:
Drug: Zinc Sulphate — 20 mg per day, Zinc Sulphate tablet has been given to subjects.
  Other Names: Zincol
  Arms: A
Drug: Zinc Sulphate — 20 mg per day of Zinc Sulphate in suspension form has been given to subjects.
  Other Names: Zincat
  Arms: B

SUMMARY:
This project is aimed to evaluate the efficacy of two different zinc formulations (dispersible Zinc tablets versus Zinc suspension) for the treatment of acute diarrhea in hospital based settings. Additionally we intend to compare the effectiveness of treatments of different groups on the basis of usage of Zinc in the treatment of diarrhoea, and to monitor additional treatment components such as ORS, antibiotic usage rates.

DETAILED DESCRIPTION:
This will be an open randomized trial in children designed to measure the impact and efficacy of daily zinc administration. There will be two groups in the study, one group will receive Zinc in the form tablets, other will receive in the form of suspension, both of these groups will also receive recommended treatment of diarrhea as per WHO protocol and these groups will be enrolled from the patients admitting in the Paediatric Unit of Civil Hospital, Hyderabad and NICH, Karachi with the complain of acute diarrhoea.

The intervention study will be undertaken in hospital based settings. A total recruitment of 300(150 each in each group) has been targetted during the study duration. The duration of this study shall be 9 months.

A brief history will be taken regarding the current illness and will be noted down in the specific forms. After the history the patient will be completely examined by the duty doctors, examination will emphasize of the vitals, status of dehydration and anthropometry. Patient will then be randomized in one of the groups and the procedure of using Zinc tablets or suspension will be explained to the mother or caretaker.The patient will be advised treatment according to the general condition and state of the dehydration and general health. All treatments will be noted down in the specific forms to have a record of what have been given to the patient and to keep the record of fluid intake. Stool samples for the detailed report and culture and sensitivity will be collected & sent to have the information regarding the status of stool and any isolated organism.

Follow-ups

* The patients will be followed & examined thoroughly every 8 hourly till the time of discharge by a trained RMO.
* At each follow up, details of illness characteristics, including the number and character of stools and vomiting, will be obtained.
* Information regarding the associated symptoms including fever, abdominal pain distension and dysentery will be obtained. Hydration status, vitals and weight will also be assessed.
* RMO will record about the proper dosages of zinc and confirm that weather or not patient is taking his medications during every follow up
* RMO will also document the recovery of diarrhea in terms of reduction in frequency and duration of diarrhoea and all the information will be noted in the assigned follow up forms.
* Any adverse effect of the associated with the Zinc will also be recorded.
* Compliance will be measured by reported intake and by measuring the remaining volume of syrup in the returned bottles and number of tablets used in the blisters.
* At the time of discharge a discharge summary form is also filled by RMO
* The patients who will be discharged will be followed at home for a total of two weeks of illness.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 months to 5 years of age
* Presented with passage of 3 or more loose or watery stools
* Caretakers are willing to let their child to participate in the study.

Exclusion Criteria:

* Failure to produce consent.
* Children with severe malnutrition or having chronic illness

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Comparison of Efficacy of the two different Zinc Sulphate formulations | 9 months

SECONDARY OUTCOMES:
Comparison of side effects of the two different Zinc Sulphate formulations used | 9 months

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Civil Hospital, Hyderābād, Sindh
  - National Institute of Child Health, Karachi, Sindh